CLINICAL TRIAL: NCT02983292
Title: A Clinical and Radiological Study to Evaluate the Safety and Efficacy of the PyroTITAN Humeral Resurfacing Arthroplasty (HRA) Device in a New Cohort of Patients After Product Re-Release
Brief Title: PyroTITAN Humeral Resurfacing Arthroplasty (HRA)
Acronym: HRA
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T-HRA-003
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-06

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PyroTITAN™ HRA — Humeral Resurfacing

SUMMARY:
The study is designed as a single center, post-market, non-randomized, open-label, observational clinical study with retrospective and prospective enrollment to evaluate the 2-year post implantation survivorship of the PyroTITAN™ HRA device following the implementation of a new proof test to identify and eliminate devices with sub-standard mechanical integrity.

DETAILED DESCRIPTION:
The study is designed as a single center, post-market, non-randomized, open-label, observational clinical study with retrospective and prospective enrollment to evaluate the 2-year post implantation survivorship of the PyroTITAN™ HRA device following the implementation of a new proof test to identify and eliminate devices with sub-standard mechanical integrity. The results will be compared to data collected in a prior study conducted before implementing the new proof test. The PyroTITAN™ HRA Shoulder prosthesis device configuration will include humeral resurfacing CAP without cement. Patients will be selected retrospectively and prospectively for recruitment into the study based upon the normally accepted criteria for primary shoulder resurfacing arthroplasty.

137 subjects with PyroTITAN™ HRA Shoulder prosthesis arthroplasties will be implanted and followed for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

Patients of either sex will be included, if they:

1. Present (prospective cohort) or presented (retrospective cohort) for primary shoulder surface replacement or arthroplasty with any of the following diagnoses:

   1. Osteoarthritis
   2. Rheumatoid / Inflammatory Arthritis
   3. Post-traumatic arthritis.
   4. Focal and large (Hill-Sachs) osteochondral defects.
2. Subject receives (prospective cohort) the PyroTITAN HRA device after the re-release of the product or received (retrospective cohort) the PyroTITAN HRA device after the re- release of the product and is enrolled in the study prior to their two-year follow-up visit.
3. Subject is able to or capable of providing consent to participate in the clinical investigation.
4. Subject agrees to comply with this protocol, including participating in required follow-up visits at the investigations site and completing study questionnaires.
5. Subject is at least 18 years of age and skeletally mature at the time of surgery.

Exclusion Criteria:

Patients will be excluded from participation if they:

1. Has/had destruction of the proximal humerus to preclude rigid fixation of the humeral component.
2. Has/had insufficient bone quality as determined by intra- operative evaluation.
3. Has/had arthritis with defective rotator cuff.
4. Has/had had a failed rotator cuff surgery.
5. Has/had loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
6. Has/had evidence of active infection.
7. Present/presented with a condition of neuromuscular compromise of the shoulder (e.g., neuropathic joints or brachioplexus injury with a flail shoulder joint).
8. Are unwilling or unable to comply with a rehabilitation program or would fail to return for the postoperative follow- up visits prescribed by the protocol.
9. Are/were skeletally immature.
10. Has/had a known allergic reaction to PyroCarbon.
11. Has/had other conditions such as central nervous system disturbances, alcohol or drug addiction, etc. that may make effective evaluation of the joint replacement difficult or impossible.
12. Has/had known, active metastatic or neoplastic disease.
13. Are/were taking > 10mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery.
14. Are/were under 21 years of age or over 75.
15. Require/required glenoid replacement.
16. Retrospective patients cannot be enrolled if they are two year or greater out from the index surgery.
17. Women, who are pregnant or are planning to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who require humeral head resurfacing arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Larson, Study Director — Smith & Nephew, Inc.
Locations (1):
- The Brisbane Hand and Upper Limb Research Institute, Brisbane, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at one (1) site in Australia and participated between 24 Oct 2016 to 08 Feb 2023.
Pre-assignment Details: Overall, 137 participants were enrolled in the study, and fifty-two (52) participants discontinued from the study before completion.
Groups:
- PyroTITAN™ HRA Shoulder System: Participants implanted with PyroTITAN™ Humeral Resurfacing Arthroplasty (HRA) Shoulder System
Period: Overall Study
Arm/Group | PyroTITAN™ HRA Shoulder System
Started | 137
Completed | 85
Not Completed | 52
Not completed — Participant unwell & cannot travel | 2
Not completed — Lost to Follow-up | 3
Not completed — Participant withdrew consent | 2
Not completed — Revision | 7
Not completed — Death | 1
Not completed — Participant did not return due to COVID-19 related lockdown | 30
Not completed — Participant failed to return for follow-up visits | 6
Not completed — Participant relocation | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population included all participants implanted with available data available.
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 137
Dominant Side [Count of Participants; unit: Participants]
  Right | 123
  Left | 14
  Missing | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Device Survival: Kaplan-Meir Estimate
Description: Device survival was defined as the absence of device fracture at the two year time-point. Percentage of participants with survival of the device estimated using the Kaplan-Meier method.
Time Frame: 2 years
Population: Participants with data available at the time frame indicated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 114
percentage of participants | 98.47 [96.35 to 100.0]

2. Secondary Outcome: Number of Participants With Device-Related Adverse Events
Description: Count of participants with device-related Non-Serious & Serious Adverse Events were the event was related to device use (e.g., component breakage) as determined by investigator assessment.
Time Frame: Post-operatively to 5-Years
Population: Participants with data available at the time frame indicated
Measure: Count of Participants; unit: Participants
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 137
Participants
  Device-Related Non-Serious Adverse Event | 6
  Device-Related Serious Adverse Event | 6

3. Secondary Outcome: Cumulative Device Success
Description: Device success was defined as the absence of device fracture over time. Cumulative device success was determined by the percentage of participants with no device fractures by the two year & five year time-points.
Time Frame: 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 118
percentage of participants
  2-Years | 98.5 [96.3 to 100.0]
  5-Years: number analyzed (Participants) | 85
  5-Years | 97.5 [94.6 to 100.0]

4. Secondary Outcome: Cumulative Device Survival
Description: Device survival was defined as the absence of device revision over time. Cumulative device survival was determined by the percentage of participants with no device revisions by the two year & five year time-points.
Time Frame: 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 118
percentage of participants
  2-Years | 96.24 [93.01 to 99.48]
  5-Years: number analyzed (Participants) | 85
  5-Years | 94.17 [89.92 to 98.42]

5. Secondary Outcome: Device Functionality: American Shoulder and Elbow Surgeons (ASES) Score
Description: ASES scores range from 0 to 100, with a score of 0 indicating a worse shoulder condition and 100 indicating the best shoulder condition.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 125
score on a scale
  Baseline | 31.1 (19.7)
  2-Years: number analyzed (Participants) | 100
  2-Years | 83.7 (18.8)
  5-Years: number analyzed (Participants) | 80
  5-Years | 88.1 (16.5)

6. Secondary Outcome: Device Functionality: Visual Analog Scale (VAS) - Pain
Description: The VAS Pain score range was from 0 to 100, with 0 representing no pain and 100 representing the worse possible pain.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 131
score on a scale
  Baseline | 66 (21)
  2-Years: number analyzed (Participants) | 112
  2-Years | 12.4 (17.4)
  5-Years: number analyzed (Participants) | 85
  5-Years | 9.5 (15.9)

7. Secondary Outcome: Device Functionality: Visual Analog Scale (VAS) - Satisfaction
Description: The VAS Satisfaction score range was from 0 to 100, with 0 representing the worst result and 100 representing the best result.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 130
score on a scale
  Baseline | 15.6 (18.5)
  2-Years: number analyzed (Participants) | 112
  2-Years | 89.6 (18.9)
  5-Years: number analyzed (Participants) | 85
  5-Years | 92.5 (13.1)

8. Secondary Outcome: Device Functionality: Western Ontario Osteoarthritis Score (WOOS)
Description: The WOOS score was based on 19 questions ranging from 0 to 100 with 0 being the best result and 100 being the worst result. A lower score indicated a better outcome.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 133
score on a scale
  Baseline | 66.7 (14.1)
  2-Years: number analyzed (Participants) | 111
  2-Years | 14.2 (89.1)
  5-Years: number analyzed (Participants) | 85
  5-Years | 11.6 (14.5)

9. Secondary Outcome: Device Functionality: QuickDASH Outcome Measure
Description: The QuickDASH (Disabilities of the Arm, Shoulder, and Hand) score ranged from 0 (no disability) to 100 (most severe disability) based on 11 questions scored 1 to 5 each (for disability/symptoms) and 4 questions scored 1 to 5 each (for performance/sport/work). A lower score indicates a better outcome.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 137
score on a scale
  Baseline | 49.5 (16)
  2-Years: number analyzed (Participants) | 110
  2-Years | 15.5 (17.1)
  5-Years: number analyzed (Participants) | 85
  5-Years | 14.5 (17)

10. Secondary Outcome: Device Functionality: Constant Murley Score (CMS)
Description: The Constant Murley Score (CMS) is a 100-point scale composed of individual parameters. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and Range of Motion (ROM) (40 points). Subscales are combined to indicate a total CMS score. The total CMS score ranges from 0 to 100 points, with higher scores indicating a better outcome.
Time Frame: Baseline, 2-Years and 5-Years
Population: Participants with data available at the time frame indicated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PyroTITAN™ HRA Shoulder System
Number analyzed (Participants) | 97
score on a scale
  Baseline: number analyzed (Participants) | 32
  Baseline | 50.7 (15)
  2-Years | 79.9 (10.3)
  5-Years: number analyzed (Participants) | 68
  5-Years | 83.7 (10.9)

ADVERSE EVENTS:
Time Frame: Surgery to end of study visit, up to 5 years
Description: All postoperative device-related & surgery-related AEs reported. Specifically, all component removals (and/or revisions) whether device related or not were recorded. Other AEs may be classified as device-related (or non device-related) based on frequency, medical significance, & circumstance. An Adverse Event Monitoring Board (AEMB), in compliance with ISO 14155 standards, classified AE relatedness as separate findings.
Arm/Group | PyroTITAN™ HRA Shoulder System
All-Cause Mortality (participants affected / at risk) | 1/137
Serious Adverse Events (participants affected / at risk) | 47/137
Other Adverse Events (participants affected / at risk) | 12/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PyroTITAN™ HRA Shoulder System (N=137)
Right shoulder rotator cuff pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Duke C Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not related to Procedure or Device
Urosepsis following surgery for prostate cancer biopsy (Surgical and medical procedures) | 1 (1) — Not related to Procedure or Device
Meniscus tear in left knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
cancerous nodule thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not related to Procedure or Device
Locking right knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Fractured left scaphoid following a fall. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
worsening OA left knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Worsening of OA in right knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Back pain exacerbated (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Deterioration of left shoulder secondary to pre-existing condition (avacular necrosis). (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Thoracic outlet syndrome progression (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Right shoulder rotator cuff impingement (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Right shoulder posterior instability (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Joint metallosis in right (operative) shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Right shoulder OA worsening (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Benign prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not related to Procedure or Device
Cardiac chest pain (Cardiac disorders) | 1 (1) — Not related to Procedure or Device
Aggravation of OA in left thumb and wrist (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Persistent right rotator cuff pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Anterior shoulder pain due to subscap impingement on the anterior aspect of the hemiarthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Fracture of PyroTITAN prosthesis. (Product Issues) | 1 (1) — Device related
Cellulitis and recurring infection in right knee (Infections and infestations) | 1 (1) — Not related to Procedure or Device
Left shoulder rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Broken right ankle (Injury, poisoning and procedural complications) | 1 (1) — Not related to Procedure or Device
Undisplaced fracture of implant (Product Issues) | 1 (1) — Device related
Worsening of OA in left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Worsening knee OA and pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Difficulty with function and ROM in left operative shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Ongoing pain in left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Right subscapular bursa irritation. (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Right shoulder full thickness tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Right leg cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Rotator cuff tendonitis left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Exacerbation of OA in right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Exacerabated right shoulder OA. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Cellulitis in left leg. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Knife injury to left arm (Injury, poisoning and procedural complications) | 1 (1) — Not related to Procedure or Device
Thoracic outlet syndrome progression. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Rotator cuff impingement left shoulder. (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
worsening osteoarthritis left wrist (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Exacerbation of OA right knee. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Subscapular bursa irritation left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Procedure Related
Fractured prosthesis (Product Issues) | 1 (1) — Device related
Worsening left shoulder osteoartritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Ongoing pain in right operative shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to Procedure or Device
worsening Osteoarthritis in right foot (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Worsening left shoulder osteoarthritis. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Worsening right shoulder arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Worsenning osteoarthritis bilateral knees. (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Pneumonia (Infections and infestations) | 1 (1) — Not related to Procedure or Device
Exacerbation of lower back nerve pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Procedure or Device
Infection left shoulder wound (Infections and infestations) | 1 (1) — Procedure Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PyroTITAN™ HRA Shoulder System (N=137)
Minor rotator cuff tendonitis left shoulder. (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Suspected stress fracture of posterior glenoid osteophyte right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Bursitis right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Squeaking right shoulder after physiotherapy. (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure or device
Cuff pain right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Suspected rotator cuff tendonitis left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not relate to procedure or device
Suspected rotator cuff tendonitis right. (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure
Crepitation around right shoulder joint with activity (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to Device
Occasional pain up right arm (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure or device
Audible squeaking left pyrotitan shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Audible squeak on flexion/extension of operative shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Persistent operative shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure or device
Skin irritation of scar in operative shoulder (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related to procedure
right shoulder stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to procedure or device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02983292/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02983292/SAP_001.pdf